CLINICAL TRIAL: NCT01940094
Title: The Assessment of Prednisone In Remission Trial (TAPIR) - Centers of Excellence Approach
Brief Title: The Assessment of Prednisone In Remission Trial - Centers of Excellence Approach
Acronym: TAPIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Principal Investigator, Peter Merkel, Chief, Division of Rheumatology, Professor of Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCRC5526A; R01HL115041 (NIH); U54AR057319 (NIH)
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Granulomatosis With Polyangiitis
Keywords: Granulomatosis with polyangiitis; Wegener's granulomatosis; WG; GPA; ANCA-Associated Vasculitis; AAV; Vasculitis; Prednisone; Glucocorticoid; Taper
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis | interventions — Prednisone; Glucocorticoids; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 mg Prednisone (Experimental): Subjects will be randomized to a prednisone dose of 5 mg per day for a 6 month period.
  Interventions: Drug: 5 mg Prednisone
- 0 mg Prednisone (Experimental): Subjects will be randomized to taper their prednisone dose from 5 mg per day to 0 mg per day for a 6 month period.
  Interventions: Drug: 0 mg Prednisone

INTERVENTIONS:
Drug: 5 mg Prednisone — Subjects will remain on daily prednisone dose of 5 mg
  Other Names: •5 mg/day glucocorticoids; •5 mg/day prednisone; •5 mg/day steroids
  Arms: 5 mg Prednisone
Drug: 0 mg Prednisone — Subjects will taper their prednisone dose from 5 mg per day to 0 mg per day
  Arms: 0 mg Prednisone

SUMMARY:
This study is a multi-center randomized controlled trial to evaluate the effects of using low-dose prednisone as compared to stopping prednisone treatment entirely. Participants will be randomized 1:1 to taper their prednisone dose down to 5 mg/day or to 0 mg/day for the duration of the study (approximately six months) or until a study endpoint.

DETAILED DESCRIPTION:
Patients with granulomatosis with polyangiitis (GPA, Wegener's) will be recruited at one of the Vasculitis Centers of Excellence. Participants will be randomized 1:1 either to taper their prednisone dose down to 5 mg/day according to a standardized schedule and stay at 5 mg/day of prednisone for the duration of the study or until a study endpoint, or taper their prednisone dose down to 0 mg/day using a standard schedule and stay at 0 mg/day for the duration of the study or until a study endpoint. All study participants will be followed for 6 months (from reaching a prednisone dose of 5 mg/day) or until an increase of prednisone dose (after randomization) occurs, whichever comes first.

Participants will have up to four study visits, a screening visit (visit 1), a baseline (visit 2), a month 3 visit (visit 3) and a month 6 or flare visit (visit 3) and up to two follow-up phone calls from the study coordinator at randomization and at month 1 (randomization and 1 month phone call may be combined if randomization occurs at month 1).

This study is a project of the Vasculitis Clinical Research Consortium (VCRC) funded through the National Institutes of Health Rare Diseases Clinical Research Network (RDCRN) with the purpose of promoting vasculitis research. The VCRC is the major clinical research infrastructure in North America for the study of vasculitis, and eight VCRC Centers of Excellence will be recruiting for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of granulomatosis with polyangiitis (GPA) where patients will need to meet at least 2 of the 5 for the classification of GPA, at least one of which must be criterion d or e:

   The modified American College of Rheumatology (ACR) criteria are:

   A. Nasal or oral inflammation, defined as the development of painful or painless oral ulcers or purulent or bloody nasal discharge.

   B. Abnormal chest radiograph, defined as the presence of nodules, fixed infiltrates, or cavities.

   C. Active urinary sediment, defined as microscopic hematuria (>5 red blood cells per high power field) or red blood cell casts.

   D. Granulomatosis inflammation on biopsy, defined as histologic changes showing granulomatous inflammation within the wall of an artery or in the perivascular or extravascular area. Note: Pauci-immune glomerulonephritis seen on kidney biopsy will suffice for this criterion.

   E. Positive anti-neutrophil cytoplasmic antibody (ANCA) test specific for proteinase-3 measures by enzyme-linked immunoassay.

   Patients who are myeloperoxidase (MPO) positive or ANCA negative are still eligible for this study if they meet the criteria above and are felt to have GPA.
2. Active disease within the prior 12 months (initial presentation or relapse) that at time of active disease required treatment with prednisone >20 mg/day.
3. Disease remission at time of enrollment.
4. Prednisone dose at time of enrollment of ≥ 5 mg/day and ≤ 20 mg/day.
5. Participant age of 18 years or greater.
6. If the patient is taking an immunosuppressive medication agent other than prednisone (maintenance agent) then the maintenance agent must be at a stable dose for one month prior to enrollment with no plans by the treating physician to change the dose (other than for safety purposes/toxicity) for the duration of the study (through the month 6 visit or early termination). Acceptable maintenance agents include azathioprine, leflunomide, 6-mercaptopurine, methotrexate, mycophenolate mofetil, mycophenolate sodium, or rituximab. Patients may be on trimethoprim/sulfamethoxazole (TMP/SMX) for use as either a maintenance agent or for prophylaxis for infection. TMP/SMX may be used in combination with other drugs.

6.1 If the patient is regularly taking trimethoprim/sulfamethoxazole at any dose then the patient is eligible if there no plans by the treating physician to change the dose after enrollment (other than dose reduction or discontinuation for safety purposes/toxicity) for the duration of the study.

Exclusion Criteria:

1. Comorbid condition that has moderate likelihood of requiring a course of prednisone within one year of enrollment (e.g. chronic obstructive pulmonary disease (COPD), asthma, adrenal insufficiency).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Physician decision to increase glucocorticoids for disease relapse. | Six months

SECONDARY OUTCOMES:
Time to disease flare. | 6 months
Safety outcomes. | 6 months
  Rate and type of serious adverse events and infections.
Protocol performance at VCRC Centers of Excellence. | 6 months
  Evaluation of patient characteristics, protocol compliance, participant retention, data completeness, timeliness of data entry, and data accuracy.
Health-related quality of life survey | Measured at baseline and end of the study
  Patient Reported Outcomes Measurement Information System (PROMIS) Assessment
Health-related quality of life surveys | Measured at baseline and the end of the study
  Measured by Short Form-36
Health-related quality of life surveys | Measured at baseline, month 3, and end of the study
  Measured by a Patient Global Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Merkel, MD, MPH, Principal Investigator — University of Pennsylvania; Jeffery P Krischer, PhD, Principal Investigator — University of South Florida
Locations (9):
- United States (7):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cronholm PF, Applequist J, Krischer J, Fontenot E, Davis T, Burroughs C, McAlear CA, Borchin R, Kullman J, Carette S, Khalidi N, Koening C, Langford CA, Monach P, Moreland L, Pagnoux C, Specks U, Sreih AG, Ytterberg SR, Merkel PA; Vasculitis Clinical Research Consortium. A study of implementation factors for a novel approach to clinical trials: constructs for consideration in the coordination of direct-to-patient online-based medical research. BMC Med Res Methodol. 2024 Oct 18;24(1):244. doi: 10.1186/s12874-024-02352-w. PMID 39425055
- See also: Vasculitis Clinical Research Consortium — http://rarediseasesnetwork.org/cms/vcrc/